CLINICAL TRIAL: NCT02322021
Title: A Placebo-Controlled, Double-Blind, Parallel-Group, Randomized, Proof-of-Concept, Dose-Finding Study To Evaluate Safety, Tolerability, and Efficacy of E2609 in Subjects With Mild Cognitive Impairment Due to Alzheimer's Disease (Prodromal Alzheimer's Disease) and Mild to Moderate Dementia Due to Alzheimer's Disease
Brief Title: Dose-Finding Study To Evaluate Safety, Tolerability, and Efficacy of E2609 in Participants With Mild Cognitive Impairment Due to Alzheimer's Disease (Prodromal Alzheimer's Disease) and Mild to Moderate Dementia Due to Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early by the sponsor on the recommendation of an independent data safety monitoring board following review of unblinded data from the Phase 3 studies E2609-G000-301 (NCT02956486) and E2609-G000-302 (NCT03036280).
Sponsor: Eisai Inc. (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2609-G000-202; 2014-002723-94 (EudraCT Number)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Alzheimer Disease; Dementia, Alzheimer Type
Keywords: E2609; Mild Cognitive Impairment; Mild to Moderate Dementia; Alzheimer's Disease; Prodromal Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- MCI/Prodromal Cohort: Low Dose (Experimental): A low dose of E2609 will be assessed.
  Interventions: Drug: E2609
- MCI/Prodromal Cohort: Middle Dose (Experimental): A middle dose of E2609 will be assessed.
  Interventions: Drug: E2609
- MCI/Prodromal Cohort: High Dose (Experimental): A high dose of E2609 will be assessed.
  Interventions: Drug: E2609
- MCI/Prodromal Cohort: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Mild to Moderate AD Cohort: Low Dose (Experimental): A low dose of E2609 will be assessed.
  Interventions: Drug: E2609
- Mild to Moderate AD Cohort: High Dose (Experimental): A high dose of E2609 will be assessed.
  Interventions: Drug: E2609
- Mild to Moderate AD Cohort: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Mild to Moderate AD cohort: Middle Dose (Experimental): A middle dose of E2609 will be assessed.
  Interventions: Drug: E2609

INTERVENTIONS:
Drug: E2609 — Each participant will receive 2 tablets, which when combined will make up the required doses of E2609 or placebo, to be administered orally once per day (QD) with food.
  Arms: MCI/Prodromal Cohort: High Dose; MCI/Prodromal Cohort: Low Dose; MCI/Prodromal Cohort: Middle Dose; Mild to Moderate AD Cohort: High Dose; Mild to Moderate AD Cohort: Low Dose; Mild to Moderate AD cohort: Middle Dose
Drug: Placebo — Each participant will receive 2 tablets, which when combined will make up the required doses of E2609 or placebo, to be administered orally once per day (QD) with food.
  Arms: MCI/Prodromal Cohort: Placebo; Mild to Moderate AD Cohort: Placebo

SUMMARY:
This is a Phase 2 study to evaluate safety and efficacy in participants with Mild Cognitive Impairment due to Alzheimer's Disease/Prodromal Alzheimer's Disease (referred to as MCI/Prodromal) and mild to moderate dementia due to Alzheimer's Disease (referred to as mild to moderate AD). This study will have a Core Phase and an Extension Phase.

ELIGIBILITY:
Inclusion criteria:

Participants must meet all of the following criteria to be included in this study:

1. Meets the core clinical research criteria of the National Institute on Aging-Alzheimer's Association (NIA-AA) for MCI due to AD (which is consistent with Prodromal AD) or AD dementia and is 'staged' or classified as either MCI or mild to moderate dementia.
2. Amyloid positive Positron Emission Tomography (PET) image based on centralized PET scan reading.
3. Male or female, age 50 to 85 years, inclusive at time of consent.
4. Must have an identified caregiver or informant who is willing and able to provide follow-up information on the participant throughout the course of the study.
5. If receiving an Acetylcholinesterase Inhibitor (AChEI) or memantine, must have been on a stable dose for at least 12 weeks before the Baseline cognitive assessments, with no plans for dose adjustment in the foreseeable future. Treatment-naive participants can be entered into the study but there should be no plans to initiate treatment with AChEIs or memantine at the time of entry into the study.
6. Must have been on stable doses of all other permitted chronically used concomitant medications (that is, not related to their cognitive decline) for at least 4 weeks before randomization.

Exclusion criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the participant's AD pathology, including any co-morbidities such as cerebrovascular disease, detected by medical history, neurological examination, or magnetic resonance imaging (MRI).
2. History of transient ischemic attacks or stroke within 12 months of Screening.
3. History of epilepsy.
4. Evidence of depression on a rating scale at Screening or any psychiatric diagnosis or symptoms, (example, hallucinations, major depression, etc.) that could confound the diagnosis or could interfere with study assessments or procedures. This includes suicidal ideation or suicidal behavior within 6 months prior to Screening, or hospitalization or treatment for suicidal behavior in the past 5 years.
5. Abnormally low serum vitamin B12.
6. Thyroid stimulating hormone above the normal range. This applies to all participants regardless of whether or not they are taking thyroid supplements.
7. Participants with liver disease (hepatic impairment), at Screening or Baseline. Participant with Gilbert's syndrome need not be excluded.
8. Not able to have a MRI, PET scanning, or cerebrospinal fluid (CSF) collection by Lumbar Puncture (LP).
9. Severe visual or hearing impairment that would prevent the participant from performing psychometric tests accurately.
10. History of immunodeficiency disorders.
11. Participants with chronic viral hepatitis.
12. History of Tuberculosis (TB). Participants with no history of TB will be tested for previous TB exposure and a positive test will be exclusionary.
13. History of ophthalmic shingles or ocular Herpes Simplex Virus (HSV) infection.
14. Any live vaccine in the 3 months or any active infection within the last 4 weeks before study drug administration (that is, randomization).
15. Any chronic inflammatory disease that is not adequately controlled or requires immunosuppressive or immunomodulatory therapy.
16. T helper cell, cytotoxic T cell, or B cell absolute counts below normal.
17. Immunoglobulin (Ig) IgG, IgA, or IgM levels below normal at Screening or Baseline, unless both the Investigator and the Medical Monitor agree that the finding is not clinically significant.
18. Clinically significant deviation from normal in physical examination, vital signs, or clinical laboratory tests at Screening or Baseline.
19. Exclusionary cardiac factors include: prolonged QT interval greater than 450 millisecond from Electrocardiograms (ECGs); history of risk factors for torsade de pointes or the use of concomitant medications that prolong the QT/corrected QT interval (QTc); left bundle branch block; persistent low or high heart rate; persistent low or high blood pressure; history of cardiac arrhythmias; other clinically significant ECG abnormalities.
20. Type 1 or Type 2 diabetes mellitus that is not well controlled.
21. Malignant neoplasms within 5 years before Screening (except for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer that did not require systemic therapy; these do not exclude the participant).
22. Medical conditions (example, cardiac, respiratory, gastrointestinal, renal disease) that are not stably controlled, or which, in the opinion of the investigator(s), could affect the participant's safety or interfere with the study assessments.
23. Hypopigmentation conditions (example, albinism and vitiligo).
24. Known or suspected history of drug or alcohol dependency or abuse within 2 years, current use of recreational drugs or a positive urine drug test.
25. Planned surgery that requires general, spinal, or epidural anesthesia that would take place during the study.
26. Participation in any other interventional clinical study related to cognitive impairment within 6 months before Screening unless it can be documented that the participant was in a placebo treatment arm.
27. Currently enrolled in another clinical study or used any investigational drug or device within 60 days or 5 half-lives of the investigational medication (whichever is longer) proceeding informed consent.
28. Hypersensitivity to the study drug or any of the excipients or to other Beta Secretase Cleaving Enzyme (BACE) inhibitors, or to the PET tracer, or components of its formulation.
29. Females who are lactating or pregnant. Females of childbearing potential who do not agree to adhere to the protocol specified methods for avoiding pregnancy.
30. Males who do not meet the protocol requirements for avoiding their partners becoming pregnant. Sperm donation is not permitted.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Bellflower, California
  - Costa Mesa, California
  - Glendale, California
  - Irvine, California
  - Aventura, Florida
  - Boca Raton, Florida
  - Brooksville, Florida
  - Lake Worth, Florida
  - Orlando, Florida
  - Port Charlotte, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Wichita, Kansas
  - Kalamazoo, Michigan
  - Mount Arlington, New Jersey
  - Scotch Plains, New Jersey
  - Charlotte, North Carolina
  - Dayton, Ohio
  - Port Royal, South Carolina
  - Dallas, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in the United States from 26 November 2014 to 20 December 2019.
Pre-assignment Details: A total of 444 participants were screened, of which 374 participants were screen failures and 70 participants were randomized and treated, out of which 43 participants completed the core phase and 41 participants entered the extension phase. No participant completed the extension phase. This study has Core Phase and an Extension Phase.
Groups:
- Core Phase: Placebo: Participants with mild cognitive impairment due to alzheimer's disease (AD)/prodromal AD and mild to moderate AD received two elenbecestat matched-placebo tablets, orally, once daily with food up to 18 months. Participants who completed 18 months treatment or who discontinued taking study drug prematurely were followed up to 3 months (12 weeks) after last dose of elenbecestat matched-placebo in core phase.
- Core Phase: Elenbecestat 5 mg Then 50 mg: Participants with mild cognitive impairment due to AD/prodromal AD and mild to moderate AD received one elenbecestat 5 milligram (mg) tablet and one elenbecestat-matched placebo tablet (to maintain blinding), orally, once daily with food up to 18 months. Participants who remained on treatment were reassigned to elenbecestat 50 mg (two 25 mg tablets) if they had at least 3 months (12 weeks) of treatment remaining in the randomization phase (treatment and follow-up), orally, once daily with food up to 18 months. Participants who completed 18 months treatment or who discontinued taking study drug prematurely were followed up to 3 months (12 weeks) after last dose of elenbecestat in core phase.
- Core Phase: Elenbecestat 15 mg Then 50 mg: Participants with mild cognitive impairment due to AD/prodromal AD and mild to moderate AD received elenbecestat 15 mg (one 10 mg and one 5 mg tablets), orally, once daily with food up to 18 months. Participants who remained on treatment were reassigned to elenbecestat 50 mg (two 25 mg tablets) if they had at least 3 months (12 weeks) of treatment remaining in the randomization phase (treatment and follow-up), orally, once daily with food up to 18 months. Participants who completed 18 months treatment or who discontinued taking study drug prematurely were followed up to 3 months (12 weeks) after last dose of elenbecestat in core phase.
- Core Phase: Elenbecestat 50 mg: Participants with mild cognitive impairment due to AD/prodromal AD and mild to moderate AD received elenbecestat 50 mg (two 25 mg tablets), orally, once daily with food up to 18 months. Participants who completed 18 months treatment or who discontinued taking study drug prematurely were followed up to 3 months (12 weeks) after last dose of elenbecestat in core phase.
- Extension Phase: Elenbecestat 50 mg: Eligible participants with mild cognitive impairment due to AD/prodromal AD and mild to moderate AD who completed the core phase entered the extension phase and received one elenbecestat 50 mg tablet, orally, once daily with or without food until early discontinuation of study drug or early termination of the study, whichever occurred first. Participants were followed up to 3 months (12 weeks) after last dose of elenbecestat in extension phase.
Period: Core Phase
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg | Extension Phase: Elenbecestat 50 mg
Started | 17 | 17 | 19 | 17 | 0
Completed | 12 | 9 | 10 | 12 | 0
Not Completed | 5 | 8 | 9 | 5 | 0
Not completed — Adverse Event | 1 | 3 | 4 | 2 | 0
Not completed — Participant Choice | 4 | 5 | 4 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg | Extension Phase: Elenbecestat 50 mg
Started | 0 | 0 | 0 | 0 | 41 (Participants who completed Core Phase, were eligible and gave consent, entered Extension Phase.)
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 41
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Participant Choice | 0 | 0 | 0 | 0 | 6
Not completed — Other | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 28

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the core phase and had at least 1 post-dose safety assessment.
Groups:
- Core Phase: Placebo: Participants with mild cognitive impairment due to AD/prodromal AD and mild to moderate AD received two elenbecestat matched-placebo tablets, orally, once daily with food up to 18 months. Participants who completed 18 months treatment or who discontinued taking study drug prematurely were followed up to 3 months (12 weeks) after last dose of elenbecestat matched-placebo in core phase.
- Core Phase: Elenbecestat 5 mg Then 50 mg: Participants with mild cognitive impairment due to AD/prodromal AD and mild to moderate AD received one elenbecestat 5 mg tablet and one elenbecestat-matched placebo tablet (to maintain blinding), orally, once daily with food up to 18 months. Participants who remained on treatment were reassigned to elenbecestat 50 mg (two 25 mg tablets) if they had at least 3 months (12 weeks) of treatment remaining in the randomization phase (treatment and follow-up), orally, once daily with food up to 18 months. Participants who completed 18 months treatment or who discontinued taking study drug prematurely were followed up to 3 months (12 weeks) after last dose of elenbecestat in core phase.
- Total: Total of all reporting groups
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg | Total
Number analyzed (Participants) | 17 | 17 | 19 | 17 | 70
Age, Customized [Count of Participants; unit: Participants]
  Less than or equal to (<=) 65 years | 4 | 3 | 2 | 3 | 12
  Greater than (>) 65 years | 13 | 14 | 17 | 14 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 12 | 10 | 42
  Male | 6 | 8 | 7 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 16 | 17 | 19 | 15 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 5 | 9
  White | 15 | 17 | 16 | 12 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an adverse event that emerges during treatment, having been absent at pre-treatment (Baseline) or re-emerges during treatment, having been present at pre-treatment (Baseline) but stopped before treatment, or worsens in severity during treatment relative to the pre-treatment state, when the adverse event is continuous.
Time Frame: Up to 21 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 17 | 17 | 19 | 17
Participants | 15 | 15 | 18 | 15

2. Primary Outcome: Core Phase: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening (that is, the participant is at immediate risk of death from the adverse event as it occurs, this does not include an event that, has it occurred in a more severe form or is allowed to continue, might have cause death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability or incapacity; is a congenital anomaly or birth defect (in the child of a participant who is exposed to the study drug).
Time Frame: Up to 21 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 17 | 17 | 19 | 17
Participants | 2 | 2 | 5 | 1

3. Primary Outcome: Core Phase: Number of Participants With Treatment Emergent Markedly Abnormal Laboratory Safety Test Values
Time Frame: Up to 21 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 17 | 17 | 19 | 17
Participants
  Markedly Abnormal Low: Lymphocytes | 0 | 2 | 0 | 0
  Markedly Abnormal Low: Leukocytes | 1 | 0 | 0 | 0
  Markedly Abnormal Low: Neutrophils | 1 | 0 | 0 | 1
  Markedly Abnormal Low: Hemoglobin | 1 | 0 | 0 | 0
  Markedly Abnormal Low: Calcium | 1 | 0 | 0 | 0
  Markedly Abnormal Low: Potassium | 0 | 0 | 1 | 0
  Markedly Abnormal High: Potassium | 2 | 4 | 2 | 0
  Markedly Abnormal High: Alkaline Phosphatase | 0 | 0 | 0 | 1
  Markedly Abnormal High: Alanine Aminotransferase | 1 | 0 | 0 | 1
  Markedly Abnormal High: Aspartate Aminotransferase | 0 | 0 | 0 | 1
  Markedly Abnormal High: Gamma Glutamyl Transferase | 1 | 0 | 0 | 1
  Markedly Abnormal Low: Glucose | 0 | 1 | 0 | 0
  Markedly Abnormal High: Glucose | 2 | 4 | 1 | 1
  Markedly Abnormal High: Cholesterol | 1 | 0 | 0 | 0
  Markedly Abnormal High: Triglycerides | 1 | 1 | 3 | 2
  Markedly Abnormal High: Creatinine | 0 | 2 | 0 | 0

4. Primary Outcome: Core Phase: Number of Participants With Markedly Abnormal Vital Sign Values
Description: Participants having no markedly abnormal vital sign values (no markedly abnormal high or no markedly abnormal low) in all core phase arms were not included in the data reported.
Time Frame: Month 0(Baseline,Week 2,Week 3,Week 4);Month 1(Week 5,Week 7);Month 2(Week 9,Week 11);Month 3(Week 13);Month 4(Week 17);Month 5(Week 21);Month 6(Week 27);Month 9(Week 40);Month 12(Week 53);Month 15(Week 66);Month 18(Week 79) and Follow-up at Month 1 and 3
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the core phase and had at least 1 post-dose safety assessment. Here "number analyzed" signifies participants who were evaluable for this outcome measure for specific categories at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 17 | 17 | 19 | 17
Participants
  Markedly Abnormal Low: Temperature (Month 0: Baseline) | 0 | 2 | 0 | 2
  Markedly Abnormal Low: Temperature (Month 0: Week 2): number analyzed (Participants) | 16 | 17 | 19 | 17
  Markedly Abnormal Low: Temperature (Month 0: Week 2) | 0 | 0 | 2 | 2
  Markedly Abnormal Low: Temperature (Month 0: Week 3): number analyzed (Participants) | 17 | 17 | 19 | 16
  Markedly Abnormal Low: Temperature (Month 0: Week 3) | 2 | 1 | 4 | 0
  Markedly Abnormal Low: Temperature (Month 0: Week 4) | 1 | 3 | 1 | 1
  Markedly Abnormal High: Temperature (Month 0: Week 4) | 0 | 0 | 1 | 0
  Markedly Abnormal Low: Temperature (Month 1: Week 5) | 1 | 0 | 2 | 0
  Markedly Abnormal Low: Temperature (Month 1: Week 7): number analyzed (Participants) | 17 | 17 | 18 | 16
  Markedly Abnormal Low: Temperature (Month 1: Week 7) | 0 | 1 | 3 | 0
  Markedly Abnormal Low: Temperature (Month 2: Week 9): number analyzed (Participants) | 17 | 17 | 15 | 16
  Markedly Abnormal Low: Temperature (Month 2: Week 9) | 0 | 1 | 1 | 2
  Markedly Abnormal Low: Temperature (Month 2: Week 11): number analyzed (Participants) | 16 | 16 | 15 | 16
  Markedly Abnormal Low: Temperature (Month 2: Week 11) | 1 | 1 | 1 | 2
  Markedly Abnormal Low: Temperature (Month 3: Week 13): number analyzed (Participants) | 16 | 16 | 15 | 16
  Markedly Abnormal Low: Temperature (Month 3: Week 13) | 1 | 2 | 3 | 1
  Markedly Abnormal Low: Temperature (Month 4: Week 17): number analyzed (Participants) | 15 | 16 | 13 | 16
  Markedly Abnormal Low: Temperature (Month 4: Week 17) | 1 | 3 | 1 | 1
  Markedly Abnormal Low: Temperature (Month 5: Week 21): number analyzed (Participants) | 15 | 16 | 13 | 16
  Markedly Abnormal Low: Temperature (Month 5: Week 21) | 1 | 3 | 0 | 0
  Markedly Abnormal Low: Temperature (Month 6: Week 27): number analyzed (Participants) | 15 | 15 | 12 | 16
  Markedly Abnormal Low: Temperature (Month 6: Week 27) | 0 | 1 | 0 | 1
  Markedly Abnormal Low: Temperature (Month 9: Week 40): number analyzed (Participants) | 14 | 13 | 11 | 15
  Markedly Abnormal Low: Temperature (Month 9: Week 40) | 1 | 2 | 0 | 1
  Markedly Abnormal Low: Temperature (Month 12: Week 53): number analyzed (Participants) | 13 | 12 | 11 | 12
  Markedly Abnormal Low: Temperature (Month 12: Week 53) | 0 | 1 | 1 | 0
  Markedly Abnormal Low: Temperature (Month 15: Week 66): number analyzed (Participants) | 13 | 11 | 10 | 12
  Markedly Abnormal Low: Temperature (Month 15: Week 66) | 0 | 3 | 2 | 2
  Markedly Abnormal Low: Temperature (Month 18: Week 79): number analyzed (Participants) | 12 | 11 | 10 | 12
  Markedly Abnormal Low: Temperature (Month 18: Week 79) | 0 | 1 | 0 | 1
  Markedly Abnormal Low: Temperature (Follow-up: Month 1): number analyzed (Participants) | 13 | 12 | 15 | 14
  Markedly Abnormal Low: Temperature (Follow-up: Month 1) | 0 | 0 | 2 | 0
  Markedly Abnormal Low: Temperature (Follow-up: Month 3): number analyzed (Participants) | 12 | 11 | 12 | 14
  Markedly Abnormal Low: Temperature (Follow-up: Month 3) | 0 | 2 | 4 | 0
  Markedly Abnormal Low: Weight (Month 0: Baseline) | 0 | 0 | 1 | 0
  Markedly Abnormal High: Weight (Month 0: Baseline) | 1 | 3 | 2 | 1
  Markedly Abnormal High: Weight (Month 3: Week 13): number analyzed (Participants) | 16 | 16 | 15 | 16
  Markedly Abnormal High: Weight (Month 3: Week 13) | 0 | 2 | 2 | 2
  Markedly Abnormal High: Weight (Month 6: Week 27): number analyzed (Participants) | 14 | 15 | 12 | 15
  Markedly Abnormal High: Weight (Month 6: Week 27) | 0 | 1 | 1 | 1
  Markedly Abnormal High: Weight (Month 9: Week 40): number analyzed (Participants) | 13 | 13 | 11 | 14
  Markedly Abnormal High: Weight (Month 9: Week 40) | 0 | 0 | 0 | 1
  Markedly Abnormal High: Weight (Follow-up: Month 3): number analyzed (Participants) | 10 | 12 | 14 | 14
  Markedly Abnormal High: Weight (Follow-up: Month 3) | 0 | 1 | 1 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 0: Baseline) | 0 | 0 | 0 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Month 0: Week 2): number analyzed (Participants) | 16 | 17 | 19 | 17
  Markedly Abnormal High: Systolic Blood Pressure (Month 0: Week 2) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 0: Week 3): number analyzed (Participants) | 17 | 17 | 19 | 16
  Markedly Abnormal High: Systolic Blood Pressure (Month 0: Week 3) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 0: Week 4) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 1: Week 5) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 1: Week 7): number analyzed (Participants) | 17 | 17 | 18 | 16
  Markedly Abnormal High: Systolic Blood Pressure (Month 1: Week 7) | 0 | 1 | 0 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 3: Week 13): number analyzed (Participants) | 16 | 16 | 15 | 16
  Markedly Abnormal High: Systolic Blood Pressure (Month 3: Week 13) | 0 | 0 | 0 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Month 4: Week 17): number analyzed (Participants) | 15 | 16 | 13 | 16
  Markedly Abnormal High: Systolic Blood Pressure (Month 4: Week 17) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Systolic Blood Pressure (Month 6: Week 27): number analyzed (Participants) | 15 | 15 | 12 | 16
  Markedly Abnormal High: Systolic Blood Pressure (Month 6: Week 27) | 0 | 0 | 1 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Month 9: Week 40): number analyzed (Participants) | 14 | 13 | 11 | 15
  Markedly Abnormal High: Systolic Blood Pressure (Month 9: Week 40) | 0 | 0 | 1 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Month 12: Week 53): number analyzed (Participants) | 13 | 12 | 11 | 12
  Markedly Abnormal High: Systolic Blood Pressure (Month 12: Week 53) | 0 | 1 | 1 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Month 15: Week 66): number analyzed (Participants) | 13 | 11 | 10 | 12
  Markedly Abnormal High: Systolic Blood Pressure (Month 15: Week 66) | 1 | 1 | 0 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Month 18: Week 79): number analyzed (Participants) | 12 | 11 | 10 | 12
  Markedly Abnormal High: Systolic Blood Pressure (Month 18: Week 79) | 0 | 1 | 1 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Follow-up: Month 1): number analyzed (Participants) | 13 | 12 | 15 | 14
  Markedly Abnormal High: Systolic Blood Pressure (Follow-up: Month 1) | 1 | 0 | 1 | 1
  Markedly Abnormal High: Systolic Blood Pressure (Follow-up: Month 3): number analyzed (Participants) | 12 | 11 | 12 | 14
  Markedly Abnormal High: Systolic Blood Pressure (Follow-up: Month 3) | 0 | 0 | 0 | 1
  Markedly Abnormal High: Diastolic Blood Pressure (Month 0: Week 3): number analyzed (Participants) | 17 | 17 | 19 | 16
  Markedly Abnormal High: Diastolic Blood Pressure (Month 0: Week 3) | 1 | 0 | 0 | 0
  Markedly Abnormal Low: Diastolic Blood Pressure (Month 0: Week 4) | 1 | 1 | 0 | 0
  Markedly Abnormal Low: Diastolic Blood Pressure (Month 1: Week 5) | 0 | 0 | 0 | 1
  Markedly Abnormal Low: Diastolic Blood Pressure (Month 9: Week 40): number analyzed (Participants) | 14 | 13 | 11 | 15
  Markedly Abnormal Low: Diastolic Blood Pressure (Month 9: Week 40) | 0 | 1 | 0 | 0
  Markedly Abnormal High: Diastolic Blood Pressure (Month 9: Week 40): number analyzed (Participants) | 14 | 13 | 11 | 15
  Markedly Abnormal High: Diastolic Blood Pressure (Month 9: Week 40) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Diastolic Blood Pressure (Follow-up: Month 1): number analyzed (Participants) | 13 | 12 | 15 | 14
  Markedly Abnormal High: Diastolic Blood Pressure (Follow-up: Month 1) | 1 | 0 | 0 | 0
  Markedly Abnormal High: Diastolic Blood Pressure (Follow-up: Month 3): number analyzed (Participants) | 12 | 11 | 12 | 14
  Markedly Abnormal High: Diastolic Blood Pressure (Follow-up: Month 3) | 0 | 0 | 0 | 1

5. Primary Outcome: Core Phase: Number of Participants With Markedly Abnormal Electrocardiogram (ECG) Findings
Description: QTcF interval means corrected QT interval (QTc) calculated using Fridericia's formula.
Time Frame: Up to 21 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 17 | 17 | 19 | 17
Participants
  At least one post-baseline increase of >30 millisecond (msec) in QTcF interval | 2 | 4 | 4 | 2
  At least one post-baseline value of >450 msec in QTcF interval | 1 | 6 | 4 | 3
  At least one post-baseline value of >480 msec in QTcF interval | 0 | 0 | 1 | 0

6. Primary Outcome: Extension Phase: Number of Participants With TEAEs and SAEs
Description: TEAE: adverse event that emerges during treatment, having been absent at pre-treatment or reemerges during treatment, having been present at pre-treatment but stopped before treatment, or worsens in severity during treatment relative to pre-treatment state. Number of participants with TEAEs were reported based on safety assessments of laboratory tests, physical examination, regular measurement of vital signs, magnetic resonance imaging and electrocardiogram parameter values. SAE: any untoward medical occurrence that at any dose: results in death; is life-threatening (immediate risk of death from adverse event, this does not include event that, had it occurred in more severe form or is allowed to continue, might have caused death); requires inpatient or prolongation of existing hospitalization; results in persistent/significant disability/incapacity; is congenital anomaly/birth defect (in child of participant exposed to drug). Number of participants with TEAEs and SAEs were reported.
Time Frame: Up to 34 months
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
Participants
  TEAEs | 30
  SAEs | 6

7. Primary Outcome: Extension Phase: Number of Participants With Markedly Abnormal Vital Sign Values
Time Frame: Up to 34 months
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
Participants
  Markedly Abnormal High: Diastolic Blood Pressure | 1
  Markedly Abnormal Low: Diastolic Blood Pressure | 1
  Markedly Abnormal High: Systolic Blood Pressure | 5
  Markedly Abnormal High: Temperature | 1
  Markedly Abnormal Low: Temperature | 10
  Markedly Abnormal High: Weight | 1

8. Primary Outcome: Extension Phase: Number of Participants With Markedly Abnormal ECG Findings
Description: QTcF interval means QTc interval calculated using Fridericia's formula.
Time Frame: Up to 34 months
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
Participants
  At least one post-baseline increase of >30 msec in QTcF interval | 2
  At least one post-baseline value of >450 msec in QTcF interval | 4

9. Primary Outcome: Extension Phase: Number of Participants With Treatment Emergent Markedly Abnormal Laboratory Safety Test Values
Time Frame: Up to 34 months
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the extension phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
Participants
  Markedly Abnormal Low: Lymphocytes | 4
  Markedly Abnormal Low: Neutrophils | 2
  Markedly Abnormal Low: Hemoglobin | 1
  Markedly Abnormal High: Potassium | 4
  Markedly Abnormal High: Alanine Aminotransferase | 1
  Markedly Abnormal High: Gamma Glutamyl Transferase | 2
  Markedly Abnormal High: Glucose | 3
  Markedly Abnormal High: Triglycerides | 2
  Markedly Abnormal High: Creatinine | 4
  Markedly Abnormal High: Urate | 1
  Markedly Abnormal Low: Platelets | 1

10. Primary Outcome: Extension Phase: Number of Participants With Abnormal Magnetic Resonance Imaging (MRI) Findings
Description: Brain MRIs are collected to assess for potential drug-related changes that might have constituted a safety concern. Safety brain MRI is assessed using a standardized procedure that included fluid-attenuated inversion recovery (FLAIR), gradient-echo, T1, and diffusion-weighted sequences to determine the presence of focal lesions including, but not limited to, evidence for ischemic and hemorrhagic stroke, subdural hematoma, neoplasm, arteriovenous malformation, micro and macrohemorrhages, superficial siderosis, lacunar infarcts, white matter abnormalities, and vasogenic edema. Participants with abnormal values related to safety brain MRI were reported.
Time Frame: Up to 34 months
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug in the extension phase. Here "number analyzed" signifies participants who were evaluable for this outcome measure for specific categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
Participants
  Brain Vasogenic Edema: number analyzed (Participants) | 27
  Brain Vasogenic Edema | 0
  Brain Microhemorrhages: number analyzed (Participants) | 23
  Brain Microhemorrhages | 4
  Brain White Matter Disease: Focal Lesions: number analyzed (Participants) | 27
  Brain White Matter Disease: Focal Lesions | 25
  Brain White Matter Disease: No Lesions: number analyzed (Participants) | 27
  Brain White Matter Disease: No Lesions | 2
  Area of superficial siderosis | 1
  Space occupying lesion (extra axial): Meningioma | 1
  Other pituitary lesion | 1

11. Secondary Outcome: Core Phase: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid (A) Beta(1-x) and Abeta(1-42) After 1 Month and 18 Months of Treatment
Description: The measurement of the amyloid proteins Abeta(1-x) and Abeta(1-42), in CSF have been shown to be important biomarkers for alzheimer's disease.
Time Frame: Month 1 (Week 5) and Month 18 (Week 79)
Population: The pharmacodynamic (PD) analysis set was the group of participants who had a baseline PD measurement and at least 1 post-dose PD measurement in the core phase. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure for specific categories and timepoints.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 4 | 7 | 6 | 6
percent change
  Percent Change from Baseline in CSF Abeta(1-x) at Month 1 (Week 5) | 6.63 (12.545) | -18.16 (17.873) | -36.43 (16.026) | -56.66 (14.431)
  Percent Change from Baseline in CSF Abeta(1-x) at Month 18 (Week 79): number analyzed (Participants) | 1 | 2 | 1 | 2
  Percent Change from Baseline in CSF Abeta(1-x) at Month 18 (Week 79) | -1.81 (NA) — Standard deviation could not be calculated due to only one participant was analyzed. | -33.86 (11.039) | -0.71 (NA) — Standard deviation could not be calculated due to only one participant was analyzed. | 33.98 (160.017)
  Percent Change from Baseline in CSF Abeta(1-42) at Month 1 (Week 5) | -8.53 (16.818) | -9.43 (22.798) | -20.69 (15.488) | -38.89 (16.378)
  Percent Change from Baseline in CSF Abeta(1-42) at Month 18 (Week 79): number analyzed (Participants) | 2 | 2 | 3 | 4
  Percent Change from Baseline in CSF Abeta(1-42) at Month 18 (Week 79) | -6.50 (24.809) | -27.19 (20.172) | -24.02 (19.949) | -56.77 (5.312)

12. Secondary Outcome: Core Phase: Mean Concentration of Elenbecestat in CSF
Time Frame: Month 1 (Week 5) and Month 18 (Week 79)
Population: The pharmacokinetic (PK) analysis set was the group of participants with at least 1 quantifiable elenbecestat plasma concentration accompanied by a documented dosing history in the core phase. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 7 | 6 | 6
nanogram per milliliter (ng/mL)
  Month 1 (Week 5) | 1.10 (0.438) | 3.71 (1.360) | 9.93 (3.568)
  Month 18 (Week 79): number analyzed (Participants) | 2 | 2 | 4
  Month 18 (Week 79) | 0.10 (0) | 2.72 (3.197) | 14.46 (3.411)

13. Secondary Outcome: Core Phase: Mean Concentration of Elenbecestat in Plasma
Time Frame: Month 0 (Week 3), Month 3 (Week 13), Month 6 (Week 27), Month 12 (Week 53): Pre-dose, 1 to 6 hours Post-dose; Month 1 (Week 5), Month 18 (Week 79): Pre-dose, 4 to 8 hours Post-dose
Population: The PK analysis set was the group of participants with at least 1 quantifiable elenbecestat plasma concentration accompanied by a documented dosing history in the core phase. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 17 | 19 | 16
ng/mL
  Month 0 (Week 3): Pre-dose: number analyzed (Participants) | 17 | 18 | 13
  Month 0 (Week 3): Pre-dose | 1.43 (1.105) | 5.81 (3.785) | 15.77 (11.281)
  Month 0 (Week 3): 1 to 6 hours Post-dose: number analyzed (Participants) | 17 | 18 | 13
  Month 0 (Week 3): 1 to 6 hours Post-dose | 4.28 (3.185) | 18.49 (11.272) | 70.41 (37.681)
  Month 1 (Week 5): Pre-dose: number analyzed (Participants) | 15 | 19 | 15
  Month 1 (Week 5): Pre-dose | 1.47 (0.870) | 6.74 (4.246) | 15.46 (10.463)
  Month 1 (Week 5): 4 to 8 hours Post-dose: number analyzed (Participants) | 16 | 19 | 16
  Month 1 (Week 5): 4 to 8 hours Post-dose | 4.80 (2.529) | 19.59 (7.940) | 66.83 (21.370)
  Month 3 (Week 13): Pre-dose: number analyzed (Participants) | 16 | 15 | 16
  Month 3 (Week 13): Pre-dose | 1.91 (1.703) | 6.90 (8.126) | 12.31 (7.007)
  Month 3 (Week 13): 1 to 6 hours Post-dose: number analyzed (Participants) | 16 | 14 | 16
  Month 3 (Week 13): 1 to 6 hours Post-dose | 6.06 (2.456) | 20.35 (8.893) | 75.15 (27.852)
  Month 6 (Week 27): Pre-dose: number analyzed (Participants) | 15 | 11 | 15
  Month 6 (Week 27): Pre-dose | 2.34 (2.196) | 9.10 (9.018) | 12.03 (8.962)
  Month 6 (Week 27): 1 to 6 hours Post-dose: number analyzed (Participants) | 15 | 12 | 15
  Month 6 (Week 27): 1 to 6 hours Post-dose | 11.11 (15.322) | 25.49 (22.247) | 71.28 (39.114)
  Month 12 (Week 53): Pre-dose: number analyzed (Participants) | 11 | 10 | 11
  Month 12 (Week 53): Pre-dose | 13.84 (18.482) | 21.03 (30.897) | 16.74 (22.804)
  Month 12 (Week 53): 1 to 6 hours Post-dose: number analyzed (Participants) | 12 | 10 | 11
  Month 12 (Week 53): 1 to 6 hours Post-dose | 49.78 (40.656) | 58.38 (65.148) | 82.55 (56.084)
  Month 18 (Week 79): Pre-dose: number analyzed (Participants) | 10 | 8 | 12
  Month 18 (Week 79): Pre-dose | 7.88 (5.896) | 7.13 (6.990) | 19.21 (13.602)
  Month 18 (Week 79): 4 to 8 hours Post-dose: number analyzed (Participants) | 9 | 8 | 11
  Month 18 (Week 79): 4 to 8 hours Post-dose | 47.16 (28.651) | 51.99 (44.656) | 70.43 (22.500)

14. Secondary Outcome: Extension Phase: Change From Extension Phase Baseline in the Mini-Mental State Examination (MMSE) Scores
Description: MMSE is a 30-point scale that measures orientation to time and place, registration, immediate and delayed recall, attention, language, and drawing. Scores ranges from 0 (most impaired) to 30 (no impairment). Lower score indicates more impairment.
Time Frame: Baseline, at Month 3, at Month 6, at Month 9, at Month 12, at Month 15, at Month 18, at Month 21, at Month 24, at Month 28 and at Month 32
Population: The full analysis set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment in the extension phase. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
score on a scale
  Baseline | 21.5 (5.67)
  Change at Month 3 | -0.6 (2.32)
  Change at Month 6: number analyzed (Participants) | 39
  Change at Month 6 | -0.6 (2.39)
  Change at Month 9: number analyzed (Participants) | 36
  Change at Month 9 | -0.9 (2.89)
  Change at Month 12: number analyzed (Participants) | 36
  Change at Month 12 | -1.4 (2.43)
  Change at Month 15: number analyzed (Participants) | 33
  Change at Month 15 | -1.8 (2.78)
  Change at Month 18: number analyzed (Participants) | 32
  Change at Month 18 | -1.7 (3.01)
  Change at Month 21: number analyzed (Participants) | 21
  Change at Month 21 | -2.5 (3.27)
  Change at Month 24: number analyzed (Participants) | 10
  Change at Month 24 | -3.9 (4.46)
  Change at Month 28: number analyzed (Participants) | 5
  Change at Month 28 | -6.4 (4.28)
  Change at Month 32: number analyzed (Participants) | 1
  Change at Month 32 | -2.0 (NA) — Standard deviation could not be calculated due to only one participant was analyzed.

15. Secondary Outcome: Extension Phase: Change From Extension Phase Baseline in the Functional Assessment Questionnaire (FAQ) Score
Description: The FAQ has 10 items concerned with performing daily tasks necessary for independent living. The caregiver or informant provides performance ratings on 10 complex activities of daily living performed within the preceding 4 weeks. Score ranges from 0 (independent) to 30 (dependent). Lower score indicates that participant can live independently. Higher score indicates that participant cannot live independently.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 41
score on a scale
  Baseline | 14.4 (7.31)
  Change at Month 3 | 1.3 (5.51)
  Change at Month 6: number analyzed (Participants) | 39
  Change at Month 6 | 1.4 (3.74)
  Change at Month 9: number analyzed (Participants) | 35
  Change at Month 9 | 2.2 (4.33)
  Change at Month 12: number analyzed (Participants) | 36
  Change at Month 12 | 2.6 (4.86)
  Change at Month 15: number analyzed (Participants) | 34
  Change at Month 15 | 3.0 (5.17)
  Change at Month 18: number analyzed (Participants) | 32
  Change at Month 18 | 3.4 (4.83)
  Change at Month 21: number analyzed (Participants) | 22
  Change at Month 21 | 3.0 (3.88)
  Change at Month 24: number analyzed (Participants) | 10
  Change at Month 24 | 6.8 (5.92)
  Change at Month 28: number analyzed (Participants) | 6
  Change at Month 28 | 9.2 (4.67)
  Change at Month 32: number analyzed (Participants) | 1
  Change at Month 32 | 15.0 (NA) — Standard deviation could not be calculated due to only one participant was analyzed.

16. Secondary Outcome: Extension Phase: Percent Change From Extension Phase Baseline in Plasma Amyloid (A) Beta(1-x) Measurements at Months 12 and 24
Description: The measurement of the amyloid protein Abeta(1-x), in plasma has been shown to be an important biomarker for alzheimer's disease.
Time Frame: Month 12 and Month 24
Population: The PD analysis set was the group of participants who had at least 1 post-treatment PD measurement in the extension phase. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. Here "number analyzed" signifies participants who were evaluable for this outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 27
percent change
  Percent Change from Extension Phase Baseline in plasma Abeta(1-x) at Month 12 | -71.8 (23.30)
  Percent Change from Extension Phase Baseline in plasma Abeta(1-x) at Month 24: number analyzed (Participants) | 5
  Percent Change from Extension Phase Baseline in plasma Abeta(1-x) at Month 24 | -71.1 (31.20)

17. Secondary Outcome: Extension Phase: Percent Change From Extension Phase Baseline in Total Hippocampal Volume at Month 24
Description: Total hippocampal volume is measured by volumetric magnetic resonance imaging (vMRI). Volumetric imaging is a 3D technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Total hippocampal volume is calculated by summing up right and left hippocampal volumes.
Time Frame: Month 24
Population: The full analysis set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment in the extension phase. Here "overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 12
percent change | -4.33 (2.080)

18. Secondary Outcome: Extension Phase: Percent Change From Extension Phase Baseline in Left and Right Hippocampal Volume at Month 24
Description: Left and right hippocampal volume is measured by vMRI. Volumetric imaging is a 3D technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Left and right hippocampal volumes represent a summary measure in the left and right hippocampal regions.
Time Frame: Month 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 12
percent change
  Percent Change at Month 24 (Left Hippocampal Volume) | -4.31 (2.065)
  Percent Change at Month 24 (Right Hippocampal Volume) | -4.37 (2.667)

19. Secondary Outcome: Extension Phase: Percent Change From Extension Phase Baseline in Whole Brain Volume at Month 24
Description: Whole brain volume is measured by vMRI. Volumetric imaging is a 3D technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Whole brain volume represents a summary measure of total brain parenchyma which includes the cerebrum, basal ganglia, diencephalon, and cerebellum.
Time Frame: Month 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 12
percent change | -3.26 (1.555)

20. Secondary Outcome: Extension Phase: Percent Change From Extension Phase Baseline in Total Ventricular Volume at Month 24
Description: Total Ventricular Volume is measured by vMRI. Volumetric imaging is a 3D technique where all the MRI signals are collected from the entire tissue sample and imaged as a whole entity, therefore providing a high signal to noise ratio. Total ventricular volume represents a summary measure of total including right and left lateral ventricles, third ventricle and fourth ventricle of brain.
Time Frame: Month 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Extension Phase: Elenbecestat 50 mg
Number analyzed (Participants) | 12
percent change | 15.18 (8.544)

ADVERSE EVENTS:
Time Frame: Up to 55 months (Core Phase: Up to 21 months; Extension Phase: Up to 34 months)
Description: Adverse events were collected for all the participants who were in the safety analysis set. The safety analysis set was the group of participants who received at least 1 dose of study drug (Core and Extension Phase) and had at least 1 post-dose safety assessment (only Core Phase).
Arm/Group | Core Phase: Placebo | Core Phase: Elenbecestat 5 mg Then 50 mg | Core Phase: Elenbecestat 15 mg Then 50 mg | Core Phase: Elenbecestat 50 mg | Extension Phase: Elenbecestat 50 mg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/19 | 0/17 | 1/41
Serious Adverse Events (participants affected / at risk) | 2/17 | 2/17 | 5/19 | 1/17 | 6/41
Other Adverse Events (participants affected / at risk) | 15/17 | 15/17 | 18/19 | 15/17 | 30/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Placebo (N=17) | Core Phase: Elenbecestat 5 mg Then 50 mg (N=17) | Core Phase: Elenbecestat 15 mg Then 50 mg (N=19) | Core Phase: Elenbecestat 50 mg (N=17) | Extension Phase: Elenbecestat 50 mg (N=41)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Affective disorder (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningoencephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Phase: Placebo (N=17) | Core Phase: Elenbecestat 5 mg Then 50 mg (N=17) | Core Phase: Elenbecestat 15 mg Then 50 mg (N=19) | Core Phase: Elenbecestat 50 mg (N=17) | Extension Phase: Elenbecestat 50 mg (N=41)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular Block Second Degree (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Valve Stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right Ventricular Enlargement (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular Rosacea (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis Microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intra-Abdominal Haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Peritoneal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Breast Complication Associated With Device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Peripheral Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (6) | 4 (4) | 1 (1) | 4 (6) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (4) | 1 (3) | 1 (1) | 3 (5)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 2 (2) | 3 (3) | 4 (5)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-Lymphocyte Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bacterial Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Calcium Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Cholesterol Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Immunoglobulin G Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Potassium Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Potassium Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood Sodium Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cd4 Lymphocytes Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cd8 Lymphocytes Decreased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Monocyte Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological Examination Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Olfactory Test Abnormal (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primitive Reflex Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Rate Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Romberg Test Positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature Perception Test Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Casts (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebellar Microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral Microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Decreased Vibratory Sense (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmetria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Superficial Siderosis Of Central Nervous System (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Vasogenic Cerebral Oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 5 (6)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Hallucination, Visual (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersexuality (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Nightmare (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rapid Eye Movement Sleep Behaviour Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thinking Abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Artery Stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Turbinate Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (3) | 3 (3) | 3 (3)
Erythematotelangiectatic Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroid Cyst (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcerative Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Propulsive Gait (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Product Administration Error (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver Function Test Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occult Blood Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic Specific Antigen Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coordination Abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postural Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia Alzheimer's Type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early by the sponsor on the recommendation of an independent data safety monitoring board following review of unblinded data from the Phase 3 studies E2609-G000-301 (NCT02956486) and E2609-G000-302 (NCT03036280).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT02322021/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT02322021/SAP_001.pdf